CLINICAL TRIAL: NCT02327364
Title: Rare Disease Clinical Research Network Natural History of Pearson Syndrome North American Mitochondrial Disease Consortium (NAMDC)
Brief Title: Natural History of Pearson Syndrome
Status: Completed | Type: Observational
Sponsor: Sumit Parikh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Sumit Parikh, Associate Professor of Neurology, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: NAMDC7408
Record Dates: First submitted 2014-12-22; First posted 2014-12-30 (Estimated); Last update posted 2025-11-03 (Actual); Status verified 2020-08

CONDITIONS: Pearson Syndrome
MeSH Terms: conditions — VLCAD deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood samples will be obtained for analyses of mtDNA deletions and hematologic parameters
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this 3-year, multi-site, non-randomized, prospective, observational study is to characterize the natural history of Pearson Syndrome. The Syndrome is a rare mitochondrial disorder due to a large-scale mtDNA deletion. Children typically present in their 1st two years of life (most in infancy) with anemia and/or pancreatitis. Most individuals with Pearson Syndrome die in childhood. Those who survive evolve to Kearns-Sayre Syndrome/Chronic Progressive External Ophthalmoplegia (KSS/CPEO) although accurate survival estimates are not yet known.

DETAILED DESCRIPTION:
All patients with confirmed Pearson Syndrome who satisfy the inclusion/exclusion criteria will be offered enrollment into this study. Patients followed at participating NAMDC clinical sites will be enrolled at those sites. Patients who are not followed at participating NAMDC clinical sites and wish to participate may contact one of the member sites directly or their local doctor may direct them to one of the member sites. Both male and female patients from all racial and ethnic backgrounds who satisfy the inclusion and exclusion criteria will be encouraged to participate. Children and adults will be eligible to be enrolled, but we expect the patient population to be mostly children.

Each patient with Pearson Syndrome who enrolls in the NAMDC Clinical Registry will be encouraged to participate in this study. Each patient enrolling in this study will be required to enroll in the NAMDC Clinical Registry either prior to or upon enrolling in this study. Demographic, medical history, biochemical, histological, genetic, and other clinical data from the registry will be incorporated into this study.

Every effort will be made to minimize the inconvenience to patients of participating in this study. The study-related activities at each patient visit will be kept to a maximum of one hour, and will, whenever possible, be scheduled to coincide with the patient's regular follow-up with his or her treating physician. This study is observational and has no associated medical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. All individuals of any age with confirmed Pearson Syndrome are eligible to participate. Pearson Syndrome requires the presence of a large-scale mtDNA deletion along with sideroblastic anemia with or without pancreatic insufficiency.
2. All patients must agree to participate in the NAMDC Clinical Registry

Exclusion Criteria:

1. Patient does not fulfill criteria for Pearson Syndrome
2. Not willing to participate in the NAMDC clinical Registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed Pearson Syndrome
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2014-03; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Track patients with Pearson Syndrome longitudinally | 3 years

SECONDARY OUTCOMES:
Determine genetic and clinical predictors of Pearson Syndrome course | 3 years